CLINICAL TRIAL: NCT02964312
Title: Spirox Latera™ Implant Support of Lateral Nasal Wall Cartilage (LATERAL-OFFICE) Study
Brief Title: LATERA-OFFICE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spirox, Inc. (Industry)
Collaborators: New Arch Consulting (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-CP-302
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Nasal Obstruction
Keywords: nasal valve collapse; absorbable nasal implant
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: Single-arm intervention with pre/post comparison for treatment response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Latera Implant (Other): Unilateral or bilateral placement of the Latera nasal implant for support of the lateral nasal wall cartilage.
  Interventions: Device: Nasal Implant

INTERVENTIONS:
Device: Nasal Implant — Latera implant placed as a standalone procedure or in conjunction with a turbinate reduction procedure in an office setting under local anesthesia.

SUMMARY:
Prospective, multicenter, nonrandomized, single-arm controlled study to obtain outcomes data in participants with severe to extreme class NOSE scores who are undergoing placement of the Spirox Latera Implant with or without concurrent turbinate reduction procedures in an office setting.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has Nasal Obstruction Symptom Evaluation (NOSE) score ≥55.
2. The subject has dynamic lateral nasal wall insufficiency as confirmed by positive modified Cottle maneuver.
3. The subject is ≥18 years of age.
4. The subject is willing and able to provide informed consent and comply with the study protocol.
5. The subject is seeking treatment for nasal airway obstruction due to nasal valve collapse (NVC) and is willing to undergo an in-office nasal implant procedure alone or with a turbinate reduction procedure.
6. The subject has appropriate nasal and facial anatomy to receive the Latera Implant.
7. The subject agrees to follow-up examinations through 12 months post operatively.
8. The subject has failed to benefit from appropriate maximal medical management [eg, nasal steroids (at least 4 weeks); antihistamines; oral decongestants; nasal strips, stents, or cones]. Failure of maximal medical management may be from lack of effectiveness or tolerability.

Exclusion Criteria:

1. The subject is having a concurrent functional endoscopic sinus surgery (FESS) or sinuplasty.
2. The subject has had rhinoplasty within the past 12 months.
3. The subject is planning to have other concurrent rhinoplasty procedure.
4. The subject is planning to have other rhinoplasty procedures or will use external dilators within 12 months after the index procedure.
5. The subject has had septoplasty and/or inferior turbinate reduction within the past 6 months.
6. The subject has, in the view of the clinician, inappropriate fixation on their nasal airway.
7. The subject plans to have any surgical or nonsurgical treatment of their nasal valve, other than the index procedure, within 12 months of the study.
8. The subject has a permanent Implant or dilator in the nasal area.
9. The subject has concomitant inflammatory or infectious skin conditions or unhealed wounds in the treatment area.
10. The subject currently has active nasal vestibulitis.
11. The subject has a history of nasal vasculitis.
12. The subject is a chronic systemic steroid or recreational intranasal drug user.
13. The subject has had a cancerous or precancerous lesion and/or has had radiation exposure in the treatment area or chemotherapy.
14. The subject has polyps or pathology (ie, septal deviation) other than turbinate hypertrophy and/or lateral wall insufficiency that would contribute to airway obstruction.
15. The subject has a history of a significant bleeding disorder(s) that would prevent healing of the treatment area post procedure.
16. The subject has a known or suspected allergy to polylactide polymer (PLA) or other absorbable materials.
17. The subject has a significant systemic disease such as poorly controlled diabetes which, in the investigator's opinion, could predispose the subject to poor wound healing.
18. The subject is currently using nasal oxygen or continuous positive airway pressure (CPAP).
19. The subject is not a candidate for procedures conducted under local anesthesia and/or managed anesthesia care (MAC) or conscious sedation.
20. Female subjects of childbearing potential, known or suspected to be pregnant, or is lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Sidle, MD, Principal Investigator — Northwestern University
Locations (9):
- United States (9):
  - Beverly Hills Aesthetic Surgical Institute, Beverly Hills, California
  - Alessi Institute For Facial Plastic Surgery, Beverly Hills, California
  - ENT Assoc. of South Florida, Boca Raton, Florida
  - The Center for Sinus, Allergy, & Sleep Wellness, Boynton Beach, Florida
  - ENT of Georgia, Atlanta, Georgia
  - Chicago Nasal & Sinus Center, Chicago, Illinois
  - Madison ENT & Facial Plastic Surgery, New York, New York
  - Collin County ENT, Frisco, Texas
  - Ogden Clinic, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sidle DM, Stolovitzky P, Ow RA, Silvers S, Matheny K, Bikhazi N, Wani M, Scurry WC, Most SP. Twelve-month outcomes of a bioabsorbable implant for in-office treatment of dynamic nasal valve collapse. Laryngoscope. 2020 May;130(5):1132-1137. doi: 10.1002/lary.28151. Epub 2019 Jun 28. PMID 31254279
- [Result] Stolovitzky P, Sidle DM, Ow RA, Nachlas NE, Most SP. A prospective study for treatment of nasal valve collapse due to lateral wall insufficiency: Outcomes using a bioabsorbable implant. Laryngoscope. 2018 Nov;128(11):2483-2489. doi: 10.1002/lary.27242. Epub 2018 May 14. PMID 29756407
- [Derived] Sidle DM, Stolovitzky P, O'Malley EM, Ow RA, Nachlas NE, Silvers S. Bioabsorbable Implant for Treatment of Nasal Valve Collapse with or without Concomitant Procedures. Facial Plast Surg. 2021 Oct;37(5):673-680. doi: 10.1055/s-0041-1726464. Epub 2021 Apr 14. PMID 33853139

RESULTS

PARTICIPANT FLOW:
Groups:
- Latera Implant: Nasal Implant
  Nasal Implant: Latera implant will be placed in stand alone procedure or in conjunction with a turbinate reduction procedure
Period: Overall Study
Arm/Group | Latera Implant
Started | 166
1-Month Follow-up | 164
3-Month Follow-up | 159
6-Month Follow-up | 152
12-Month Follow-up | 139
18-Month Follow-up (The 18-mo and 24-mo follow-up visits required participants to sign an new consent to participate.) | 112
24-Month Follow-up | 102
Completed | 102
Not Completed | 64
Not completed — Lost to Follow-up | 28
Not completed — Withdrawal by Subject | 11
Not completed — Lack of Efficacy | 10
Not completed — Did not consent to long-term FU | 14
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled and treated with the Latera Implant.
Arm/Group | Latera Implant
Number analyzed (Participants) | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 84
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1
  Race: Asian | 3
  Race: Black or African American | 3
  Race: Hispanic or Latino | 11
  Race: White | 143
  Race: Other | 4
  Race: Not Specified | 1
Region of Enrollment [Number; unit: participants]
  United States | 166
NOSE score (100-point scale) [Mean (Standard Deviation); unit: units on a scale] — Nasal symptoms were evaluated using the Nasal Obstruction Symptom Evaluation (NOSE) score, a patient-reported questionnaire. The NOSE score involves rating the severity of 5 nasal symptoms (congestion, obstruction, trouble breathing, sleeping, and exercise) on a scale of 0 to 4. The values are totaled and multiplied by 5 to provide a scale of 0-100 with higher scores indicating worse symptoms.
  units on a scale | 77.4 (13.4)
Nose Severity Class [Count of Participants; unit: Participants] — NOSE severity classes are defined as Mild (5-25), Moderate (30-50), Severe (55-75), and Extreme (80-100).
  Participants
    Severe | 90
    Extreme | 76
Nasal Obstruction Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — Patient-reported instrument used to capture the participants' perception of their ability to breathe through the nose. The VAS consists of a 100-mm horizontal line marked in 1-mm increments with 0-mm indicating "no difficulty breathing through the nose" and 100-mm indicating "unable to breathe through the nose". The participant marks the point on the line that indicates their current perception.
  units on a scale | 68.0 (18.0)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percent of Treatment Responders
Description: A responder is defined as a participant who has an improvement of at least 1 NOSE class or a NOSE score reduction of at least 20% compared with baseline. NOSE scores can range from 0 to 100 with higher scores indicating worse symptoms. Classes are mild (5-25), moderate (30-50), severe (55-75) and extreme (80-100).
Time Frame: 6 months
Population: All participants who had placement of 1 or more Latera implants and had a 6-month NOSE score.
Measure: Count of Participants; unit: Participants
Groups:
- Latera Implant: Latera implant placed as a standalone procedure or in conjunction with a turbinate reduction procedure.
Arm/Group | Latera Implant
Number analyzed (Participants) | 152
Participants | 136
Statistical Analysis 1: Comparison: Latera Implant; The null hypothesis was that the proportion of responders at 6 months would be 50%. Since there was not direct comparison group, the hypothesis was set as a superiority comparison to a target proportion (66%) with a power level >90%; Test type: Superiority; Proportion = 89.5, 95% CI 2-sided [83.5 to 93.9]

2. Primary Outcome: Safety: Procedure- and/or Device-related Adverse Events
Description: Number of participants with 1 or more adverse events that are determined to be related to the Latera implant and/or procedure.
Time Frame: 6 months
Population: All participants who received 1 or more Latera implants.
Measure: Count of Participants; unit: Participants
Arm/Group | Latera Implant
Number analyzed (Participants) | 166
Participants | 31

3. Secondary Outcome: Percent of Treatment Responders
Description: as for outcome 1
Time Frame: 1, 3, 12, 18, and 24 months post procedure.
Population: All participants with NOSE scores at the applicable visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Latera Implant
Number analyzed (Participants) | 164
Participants
  1-Month Follow-up | 147
  3-Month Follow-up: number analyzed (Participants) | 156
  3-Month Follow-up | 143
  12-Month Follow-up: number analyzed (Participants) | 139
  12-Month Follow-up | 124
  18-Month Follow-up: number analyzed (Participants) | 112
  18-Month Follow-up | 103
  24-Month Follow-up: number analyzed (Participants) | 102
  24-Month Follow-up | 93

4. Secondary Outcome: Change in Nasal Airway Obstruction From Baseline Using a Visual Analog Scale (VAS)
Description: Change from baseline in the nasal obstryction VAS score. Participants provide scores on a scale of 0 (easy to breathe through the nose) to 100 (difficult to breathe through the nose) using a 100-mm line with 1-mm increments). Negative values indicate improvement in symptoms.
Time Frame: 1, 3, 6, 12, 18, and 24 months post procedure
Population: All participants with VAS scores at the applicable visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Latera Implant
Number analyzed (Participants) | 164
score on a scale
  1-Month Follow-up | -34.3 (27.0)
  3-Month Follow-up: number analyzed (Participants) | 156
  3-Month Follow-up | -35.5 (28.5)
  6-Month Follow-up: number analyzed (Participants) | 151
  6-Month Follow-up | -36.9 (29.0)
  12-Month Follow-up: number analyzed (Participants) | 139
  12-Month Follow-up | -37.9 (29.8)
  18-Month Follow-up: number analyzed (Participants) | 112
  18-Month Follow-up | -41.5 (27.3)
  24-Month Follow-up: number analyzed (Participants) | 102
  24-Month Follow-up | -41.7 (26.8)
Statistical Analysis 1: Comparison: Latera Implant; Test type: Superiority; p < 0.001, t-test, 2 sided — P values are based on paired t-tests for change from baseline with p<0.05 indicating significance

5. Secondary Outcome: Subject Satisfaction Questionnaire
Description: Participants rate whether they are satisfied or not satisfied with the procedure and cosmetic appearance after the procedure. The percent of participants reporting satisfaction with the procedure is reported.
Time Frame: 6 months
Population: All participants who completed a satisfaction questionnaire at the 6-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Latera Implant
Number analyzed (Participants) | 149
Participants | 115

6. Secondary Outcome: Procedure and Device-related Adverse Events
Description: Number of participants who experience procedure- or device-related adverse events.
Time Frame: After 6 months and up to 12 months post procedure
Population: All participants with greater than 6-months follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Latera Implant
Number analyzed (Participants) | 139
Participants | 3

ADVERSE EVENTS:
Time Frame: 24 months post procedure
Description: Participants were queried about possible adverse events at each follow-up visit. Adverse event data were collected on standardized case report forms.
Arm/Group | Latera Implant
All-Cause Mortality (participants affected / at risk) | 1/166
Serious Adverse Events (participants affected / at risk) | 0/166
Other Adverse Events (participants affected / at risk) | 24/166
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Latera Implant (N=166)
Implant migration/retrieval (Surgical and medical procedures) | 15 (16)
Sinus infection (Infections and infestations) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT02964312/Prot_SAP_000.pdf